CLINICAL TRIAL: NCT02867059
Title: A Proof-of-concept Study to Assess the Effect of (+)-SJ000557733 (SJ733) Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Participants
Brief Title: SJ733 Induced Blood Stage Malaria Challenge Study
Acronym: SJ733IBSMCS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: QIMR Berghofer Medical Research Institute (Other); Q-Pharm Pty Limited (Industry); Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QP15C20
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — SJ733

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- first dose (Experimental): The dose used in the first cohort was determined on the basis of the safety and PK data generated in the FIM study (NCT02661373) currently ongoing in United States (US) and will be 150 mg.
  Interventions: Drug: (+)-SJ000557733
- second dose (Experimental): Depending on the pharmacodynamics data (effect of SJ733 on parasitaemia) obtained from this first cohort, the dose in Cohort 2 may be adjusted but will not exceed 600 mg.
  Interventions: Drug: (+)-SJ000557733

INTERVENTIONS:
Drug: (+)-SJ000557733 — (+)-SJ000557733 (SJ733), in short SJ733, will be the second PfATP4 inhibitor to enter clinical development after KAE609 (Novartis) which is currently in Phase 2 stage. KAE609 (cipargamin; previously known as NITD609) is a spirotetrahydro-β-carbolines (spiroindolone). KAE609 inhibits QP15C20_SJ733_Challenge Protocol_v2.0_26July2016 Page 28 of 110 PfATP4, which results in a disruption of parasite sodium homeostasis. Compared to KAE609, SJ733 has the potential to be a very fast acting, antimalarial drug for human therapeutic application and may have a different safety profile in human participants. Finally, SJ733 blocks parasite transmission in vivo at potencies close to those where it is efficacious in blood stages, indicating its potential for transmission blockade in humans.
  Other Names: SJ733

SUMMARY:
This is a single-centre, open-label, study using induced blood stage malaria (IBSM) infection to characterize the activity of (+)-SJ000557733 or SJ733 for short, against early Plasmodium falciparum blood stage infection. The study will be conducted in two cohorts (n=8 per cohort). The anticipated efficacious dose range is expected to be within a range of 125 to 600 mg. The dose used in the first cohort was determined on the basis of the safety and PK data generated in the FIM study (NCT02661373) currently ongoing in United States (US) and will be 150 mg. Depending on the pharmacodynamics data (effect of SJ733 on parasitaemia) obtained from this first cohort, the dose in Cohort 2 may be adjusted but will not exceed 600 mg. Based on the PK from all three cohort from the FIM study, the median estimated dose to obtain the target SJ733 AUC of 13,000 (ug hr/L) is 370 mg. The dose of cohort 2 (≤600mg) is intended to provide further concentration-response information in the human challenge model.

For Cohort 2 only, a second dose of SJ733 may be administered at peak gametocytaemia to assess if SJ733 can reduce gametocytes and subsequent infectivity to mosquitoes (a washout of ~15 days post initial SJ733 treatment will be observed). Depending on the data obtained from the first two cohorts, there may be a subsequent cohort, with the investigated dose of SJ733 to be determined by the Sponsor and Principal Investigator (PI) and endorsed by the Safety Review Team. Should this third dose be investigated, a substantial amendment including preliminary data from the first two cohorts will be submitted to the HREC for approval.

DETAILED DESCRIPTION:
Each participant in the cohort will be inoculated on Day 0 with ~2,800 viable Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. On an outpatient basis, participants will be monitored daily via phone call and then will attend the clinic daily (AM) from day 4 (until PCR positive for presence of malaria parasites). Once PCR positive they will be monitored twice-daily, morning (AM) and evening (PM) until treatment, for adverse events and the unexpected early onset of symptoms, signs or parasitological evidence of malaria. Microscopic examination for evidence of parasitaemia may be conducted at the discretion of the Investigator. On the day designated for commencement of treatment, as determined by qPCR results, participants will be admitted to the study unit and monitored. The threshold for commencement of treatment will be when PCR quantification of all participants is ≥ 5,000 parasites/mL. If the PCR quantification of any participant is ≥ 5,000 parasites/mL, and is accompanied by a clinical symptom score >6, before all participants have reached the treatment threshold (PCR quantification of ≥ 5,000), then treatment of that participant will begin within a 24 h period.

Following treatment with SJ733, participants will be followed up as inpatients for at least 72 hours to ensure tolerance of the treatment and clinical response, then on an outpatient basis if clinically well, for monitoring of safety and clearance of malaria parasites via PCR. The plasma concentration-time profiles of SJ733 will be assessed from blood samples collected pre-dose and then following administration of the treatment drug. Wherever possible, PK sampling will coincide with post-dose blood collection for PCR monitoring of parasitaemia.

Participants may also be evaluated for the presence of gametocytes in the blood, as determined by qPCR (amplification of pfs25 gametocyte-specific transcript). Transmission blocking activity of SJ733 in P. falciparum IBSM infection may be assessed if there are >500 parasites/ml (determined by 18S qPCR) verified as gametocytes by PCR for pfs25 and/or ring stage marker as appropriate. Transmission studies may be undertaken by direct skin feeding and/or indirect membrane feeding of mosquitoes. For indirect Membrane Feeding Assays (MFA), blood will be collected from each participant for membrane feeds using Anopheles vector mosquitoes. For direct skin feeding assays (DFA), participants will be escorted to the PC3 quarantine insectary facility at QIMR Berghofer Medical Research Institute and asked to allow Anopheles vector mosquitoes to feed on the volar surface of their forearms, calves or thighs for a period of 15±5 minutes. Microscopic examination for confirmation of gametocytaemia may be conducted at the discretion of the Investigator.

If gametocytaemia is detected, in Cohort 2 only, a second same strength dose of SJ733 may be administered on Day 23, to assess if SJ733 can reduce gametocytes and subsequent infectivity to mosquitoes. To receive the second SJ733 dose, participants will have >500 parasites/ml (determined by 18S qPCR) verified as gametocytes by PCR for pfs25 and/or ring stage marker as appropriate. Membrane feeding and direct skin feeding may occur before and/or after this second SJ733 dose. Participants receiving the second SJ733 dose will visit the study unit on the morning of Day 23 for dosing and will be allowed to leave after ~10 hours. Participants will have blood samples taken during this visit at time-points indicated in the protocol.

Compulsory commencement of treatment with Riamet® (artemether-lumefantrine) will occur 16 days (±3 days) post initial SJ733 treatment unless required earlier (Cohort 1 and Cohort 2 if not given second SJ733 dose). If a second dose of SJ733 is given in Cohort 2, Riamet® treatment will occur 11 days (± 3 days) post the second SJ733 treatment unless required earlier. Early intervention can occur if either poor responses or fast responses are seen following SJ733 treatment. This is to ensure participant safety and to avoid participant inconvenience if useful data cannot be obtained. A poor response is defined as a decrease in parasitaemia of less than 20% from baseline by 3 days post SJ733 treatment. A fast response occurs when, within the seven day period, two consecutive PCR assessments in 48 hours are negative. However, pre-emptive treatment with Riamet® can commence whenever deemed necessary by the Investigator. Participants can be administered the curative Riamet® on site for initial dosing followed by monitoring, either in clinic, or by telephone for three days to ensure adherence to Riamet® therapy.

Participants will be treated with a single dose (45 mg) of primaquine (Primacin™) as described in Section 4.3 in this protocol at the time of their Riamet® treatment if gametocytes are identified, to ensure complete clearance of any gametocytes present.

Adverse events will be monitored via telephone monitoring, during confinement within the clinical research unit, and on outpatient review following malaria challenge inoculation and administration of the antimalarial treatment. Blood samples for safety evaluation, including for LFT assessment, malaria monitoring, pharmacokinetic determination of drug levels in plasma and/or blood, and red blood cell antibodies will be drawn at screening and/or baseline and at nominated times after malaria challenge.

This study includes evaluation of optional, exploratory markers, which require separate informed consent for participants agreeing to participate in any of these.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male and women of non-child bearing potential (WNCBP as defined in Section 6.17), participants between 18 and 55 years of age inclusive, who do not live alone (from Day 0 until at least the end of the antimalarial drug treatment) and will be contactable and available for the duration of the trial (maximum of 6 weeks).
* Body weight minimum 50.0 kg, body mass index between 18.0 and 32.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 5 minutes resting in supine position:

  90 mmHg ≤ systolic blood pressure (SBP) ≤ 140 mmHg, 50 mmHg ≤ diastolic blood pressure (DBP) ≤ 90 mmHg, 40 bpm ≤ heart rate (HR) ≤ 100 bpm.
* Normal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position; QTcF≤450 ms with absence of second or third degree atrioventricular block or abnormal T wave morphology.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants enrolled in this clinical investigation in accordance with Sponsor-approved clinically acceptable laboratory ranges documented prior to study start. More specifically for serum creatinine, hepatic transaminase enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the Participant has documented Gilbert syndrome) should not exceed the acceptable ranges approved by the Sponsor and haemoglobin must be equal or higher than the lower limit of the normal range.
* Male participants must agree to use a double barrier method of contraception including condom plus diaphragm or condom plus IUD or condom plus stable oral/transdermal/injectable hormonal contraceptive by female partner for at least 7 days prior to the time of the first dose of study drug through 90 days after the 5th half-life of the last dose of study drug (half-life of ~20 hours). Abstinent participants have to agree starting a double barrier method if they start sexual relationships during the study and up to 95 days after the last dose of study drug.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Any history of malaria or participation to a previous malaria challenge study.
* Must not have travelled to or lived (>2 weeks) in a malaria-endemic region during the past 12 months or planned travel to a malaria-endemic region during the course of the study (for endemic regions see http://www.map.ox.ac.uk/browse-resources/).
* Has evidence of increased cardiovascular disease risk (defined as >10%, 5 year risk for those greater than 35 years of age), as determined by the Australian Absolute Cardiovascular Disease Risk Calculator (http://www.cvdcheck.org.au/). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, total and HDL cholesterol (mmol/L) and reported diabetes status.
* History of splenectomy.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin-dependent and non-insulin dependent diabetes (excluding glucose intolerance if E03 is met), progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma.
* History of photosensitivity.
* History of G6PD deficiency.
* Participants with history of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis, including depression or receiving psychiatric drugs or who has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Migraine, recurrent nausea, and/or vomiting (more than twice a month).
* Presence of acute infectious disease or fever (e.g., sub-lingual temperature ≥ 38.5°C) within the five days prior to inoculation with malaria parasites.
* Evidence of acute illness within the four weeks before trial prior to screening that the Investigator deems may compromise participant safety.
* Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
* Participant has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhea.
* Participation in any investigational product study within the 12 weeks preceding the study.
* Participation in any research study involving blood sampling (more than 450 mL/ unit of blood), or blood donation to Red Cross (or other) blood bank during the 8 weeks preceding the treatment drug dose in the study.
* Participant unwilling to defer blood donations to the ARCBS for 6 months.
* Medical requirement for intravenous immunoglobulin or blood transfusions.
* Participant who has ever received a blood transfusion.
* Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 minutes when changing from supine to standing position.
* History or presence of alcohol abuse (alcohol consumption more than 40 g per day) or drug habituation, or any prior intravenous usage of an illicit substance.
* Tobacco use of more than 5 cigarettes or equivalent per day and unable to stop smoking during the study.
* Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (participants will be advised by phone not to consume any poppy seeds in this time period).
* Excessive consumption of beverages containing xanthine bases, including red bull, chocolate etc. more than 400 mg of caffeine per day (more than 4 cups or glasses per day).
* Any vaccination within the last 28 days.
* Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants. Any participant currently receiving or having previously received immunosuppressive therapy, including systemic steroids including adrenocorticotrophic hormone (ACTH) or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression such as 1 mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids (budesonide 800 micrograms per day or fluticasone 750 micrograms).
* Any recent (less than 6 weeks) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (chloroquine, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, hydroxychloroquine, etc.).
* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any participant in the exclusion period of a previous study according to applicable regulations.
* Any participant who lives alone (from Day 0 until at least the end of the antimalarial drug treatment).
* Any participant who cannot be contacted in case of emergency for the duration of the trial and up to 2 weeks following end of study visit.
* Any employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child whether biological or legally adopted.
* Any participant without a good peripheral venous access.Male participant with a female partner who is pregnant or lactating from the time of administration of study medication.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
* A positive urine drug test at screening, pre-inoculation, or pre any SJ733 dose. Any drug listed in Table 2 (Drug Screening) in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug) and/or the Participant has a negative urine drug screen on retest by the pathology laboratory.
* A positive alcohol breath test at screening, pre-inoculation or pre any SJ733 dose.
* Cardiac/QT risk:
* Known pre-existing prolongation of the QTcB/QTcF interval considered clinically significant.
* History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia. Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia or hypomagnesaemia.
* Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analysis.
* A history of clinically significant ECG abnormalities.
* Known hypersensitivity to SJ733 or any of its excipients or artemether or other artemisinin derivatives, lumefantrine, or other arylaminoalcohols.
* Unwillingness to abstain from consumption of citrus (grapefruit, Seville orange, etc.) for at least 28 days prior to initiation of the study (inoculation, Day 0) and for the study duration.
* Unwillingness to abstain from consumption of quinine containing foods/beverages such as tonic water, lemon bitter, from inoculation (Day 0) to the end of the antimalarial treatment.
* Use of prescription or non-prescription drugs and herbal supplements (such as St John's Wort) within 14 days or 5 half-lives (whichever is the longer) prior to the inoculation administration. (As an exception, ibuprofen (preferred) may be used at doses of up to 1.2 g/day, or paracetamol at doses of up to 2 g/day. Limited use of other non-prescription medications or dietary supplements not believed to affect subject safety or the overall results of the study, may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the Investigator.) (Note: diazepam interferes with the analysis of blood levels of SJ733 and thus should not have been used for at least 8 weeks prior to administration of the study drug).
* Known severe reaction to mosquito bites other than local itching and redness. Participants are requested to refrain from taking non-approved concomitant medication from recruitment until the conclusion of the study.

Participants who are excluded from participation on study days for any of the above reasons may be eligible to participate on a postponed schedule if the Investigator considers this appropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Q-Pharm Clinics, Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Q-Pharm Clinics, Herston, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodford J, Gillman A, Jenvey P, Roberts J, Woolley S, Barber BE, Fernandez M, Rose S, Thomas P, Anstey NM, McCarthy JS. Positron emission tomography and magnetic resonance imaging in experimental human malaria to identify organ-specific changes in morphology and glucose metabolism: A prospective cohort study. PLoS Med. 2021 May 26;18(5):e1003567. doi: 10.1371/journal.pmed.1003567. eCollection 2021 May. PMID 34038421
- [Derived] Gaur AH, McCarthy JS, Panetta JC, Dallas RH, Woodford J, Tang L, Smith AM, Stewart TB, Branum KC, Freeman BB 3rd, Patel ND, John E, Chalon S, Ost S, Heine RN, Richardson JL, Christensen R, Flynn PM, Van Gessel Y, Mitasev B, Mohrle JJ, Gusovsky F, Bebrevska L, Guy RK. Safety, tolerability, pharmacokinetics, and antimalarial efficacy of a novel Plasmodium falciparum ATP4 inhibitor SJ733: a first-in-human and induced blood-stage malaria phase 1a/b trial. Lancet Infect Dis. 2020 Aug;20(8):964-975. doi: 10.1016/S1473-3099(19)30611-5. Epub 2020 Apr 8. PMID 32275867

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Dose | Second Dose
Started | 7 | 10
Completed | 7 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Dose | Second Dose | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.14 (4.807) | 25.08 (3.261) | 25.11 (3.827)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.14 (4.807) | 25.08 (3.261) | 25.11 (3.827)

OUTCOME MEASURES:

1. Primary Outcome: Activity of SJ733 Administered Orally on Clearance of P. Falciparum Blood Stage Parasites From the Blood in Healthy Subjects (Men and WNCBP)
Description: The parasite reduction ratio (PRR) provides an estimate of the efficacy of an antimalarial treatment and is the ratio of the parasite density between admission and 48 h post antimalarial treatment. The primary efficacy variable is parasite reduction ratio (PRR) of parasites based on qPCR after administration of SJ733. The PRR was estimated using the slope of the optimal fit of the log-linear relationship of the parasitaemia decay.
  PRR was calculated for each subject using the retrospective 18S rRNA qPCR data. If the model fit was adequate for the subject (defined as overall model p-value <0.001), the slope and corresponding standard error from the log-linear regression was used to calculate the overall cohort specific PRR.
Time Frame: Until End of Study (Day 28±3)
Population: Two subjects in Cohort 2a were excluded from PRR analyses because they were not dosed with SJ733. Of the remaining 8 subjects in cohorts 2a/2b, one subject did not have a significant optimal regression fit and was excluded from the cohort-specific analysis. As such, 7 subjects contributed to calculations of a cohort-specific PRR for cohorts 2a/2b.
Measure: Mean (95% Confidence Interval); unit: Parasite Reduction Rate (PRR)
Groups:
- First Dose 150mg: The dose used in the first cohort was determined on the basis of the safety and PK data generated in the FIM study (NCT02661373) currently ongoing in United States (US) and will be 150 mg.
  (+)-SJ000557733: (+)-SJ000557733 (SJ733), in short SJ733, will be the second PfATP4 inhibitor to enter clinical development after KAE609 (Novartis) which is currently in Phase 2 stage. KAE609 (cipargamin; previously known as NITD609) is a spirotetrahydro-β-carbolines (spiroindolone). KAE609 inhibits QP15C20_SJ733_Challenge Protocol_v2.0_26July2016 Page 28 of 110 PfATP4, which results in a disruption of parasite sodium homeostasis. Compared to KAE609, SJ733 has the potential to be a very fast acting, antimalarial drug for human therapeutic application and may have a different safety profile in human participants. Finally, SJ733 blocks parasite transmission in vivo at potencies close to those where it is efficacious in blood stages, indicating its potential for transmission blockade in humans.
- Second Dose 600mg: Depending on the pharmacodynamics data (effect of SJ733 on parasitaemia) obtained from this first cohort, the dose in Cohort 2 may be adjusted but will not exceed 600 mg.
  (+)-SJ000557733: (+)-SJ000557733 (SJ733), in short SJ733, will be the second PfATP4 inhibitor to enter clinical development after KAE609 (Novartis) which is currently in Phase 2 stage. KAE609 (cipargamin; previously known as NITD609) is a spirotetrahydro-β-carbolines (spiroindolone). KAE609 inhibits QP15C20_SJ733_Challenge Protocol_v2.0_26July2016 Page 28 of 110 PfATP4, which results in a disruption of parasite sodium homeostasis. Compared to KAE609, SJ733 has the potential to be a very fast acting, antimalarial drug for human therapeutic application and may have a different safety profile in human participants. Finally, SJ733 blocks parasite transmission in vivo at potencies close to those where it is efficacious in blood stages, indicating its potential for transmission blockade in humans.
Arm/Group | First Dose 150mg | Second Dose 600mg
Number analyzed (Participants) | 7 | 7
Parasite Reduction Rate (PRR) | 172 [103 to 286] | 11551 [5348 to 24944]

2. Primary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of SJ733 in healthy subjects (men and WNCBP) following infection with blood stage P. falciparum during the IBSM challenge study will be evaluated by observation of occurrence of adverse events.
Time Frame: for up to 25th day post SJ733 treatment or longer as determind by the principal investigator
Measure: Count of Participants; unit: Participants
Arm/Group | First Dose 150mg | Second Dose 600mg
Number analyzed (Participants) | 7 | 8
Participants | 7 | 8

ADVERSE EVENTS:
Arm/Group | First Dose | Second Dose
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Dose (N=7) | Second Dose (N=8)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 6 (6) | 5 (6)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 4 (4) | 3 (3)
Puncture site erythema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (18) | 5 (9)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Urine output increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (7)
Headache (Nervous system disorders) | 6 (11) | 6 (15)
Lethargy (Nervous system disorders) | 2 (2) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days